CLINICAL TRIAL: NCT03034096
Title: General Anesthetics in CAncer REsection Surgery (GA-CARES) Trial: Pragmatic Randomized Trial of Propofol vs Volatile Inhalational Anesthesia
Brief Title: General Anesthetics in CAncer REsection Surgery (GA-CARES) Trial
Acronym: GA-CARES
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Elliott Bennett-Guerrero, Professor and Vice Chairman, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 967670-3
Record Dates: First submitted 2017-01-22; First posted 2017-01-27 (Estimated); Last update posted 2025-05-04 (Actual); Status verified 2025-01

CONDITIONS: Anesthesia, General; Surgical Oncology
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propofol infusion (Experimental): Maintenance of general anesthesia with propofol infusion
  Interventions: Drug: Propofol
- Volatile agent (Experimental): Maintenance of general anesthesia with volatile agent (sevoflurane, desflurane, or isoflurane)
  Interventions: Drug: Volatile Agent

INTERVENTIONS:
Drug: Propofol — Maintenance of general anesthesia with propofol infusion
  Arms: Propofol infusion
Drug: Volatile Agent — Maintenance of general anesthesia with volatile agent (sevoflurane, desflurane, or isoflurane)
  Arms: Volatile agent

SUMMARY:
This is a large pragmatic multicenter trial comparing maintenance of general anesthesia with total intravenous anesthesia using propofol versus volatile agent (sevoflurane, isoflurane, or desflurane) during cancer surgery. The primary endpoint is all-cause mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known or suspected cancer and scheduled to undergo any of the following oncologic surgical procedures:

  * Lobectomy or pneumonectomy
  * Esophagectomy
  * Radical (total) cystectomy
  * Pancreatectomy
  * Partial hepatectomy
  * Hyperthermic intraperitoneal chemotherapy (HIPEC)
  * Gastrectomy (subtotal or total)
  * Cholecystectomy or bile duct resection

Exclusion Criteria:

* Age less than 18 years
* American Society of Anesthesiologist Class 5
* Projected life expectancy less than 30 days
* Known or suspected hypersensitivity to either propofol, e.g. egg or soy allergy, or volatile general anesthetic agents
* Known or suspected history of malignant hyperthermia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1826 (Actual)
Dates: Start 2017-01-31 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
All-cause mortality | 2 year minimum
  Time to event

SECONDARY OUTCOMES:
Recurrence free survival | Minimum 2 years
  Time to event
All-cause mortality as a binary outcome | 2 years

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Roswell Park Cancer Center, Buffalo, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Stony Brook University Hospital, Stony Brook, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bennett-Guerrero E, Romeiser JL, DeMaria S, Nadler JW, Quinn TD, Ponnappan SK, Wang R, Gloff MS, Lee KJ, Levin MA, Sroka RD, Stanley SL, Wang D, Sasson AR; GA-CARES Trial Group. Anesthesia Type during Cancer Surgery: Results of the GA-CARES Randomized, Multicenter Trial. Anesthesiology. 2026 Jan 1;144(1):51-62. doi: 10.1097/ALN.0000000000005769. Epub 2025 Dec 9. PMID 41363871
- [Derived] Bennett-Guerrero E, Romeiser JL, DeMaria S, Nadler JW, Quinn TD, Ponnappan SK, Yang J, Sasson AR. General Anesthetics in CAncer REsection Surgery (GA-CARES) randomized multicenter trial of propofol vs volatile inhalational anesthesia: protocol description. Perioper Med (Lond). 2023 Jan 11;12(1):2. doi: 10.1186/s13741-022-00290-z. PMID 36631831